CLINICAL TRIAL: NCT01994837
Title: A Phase 2 Study of ABT-199 in Subjects With Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-212
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-01

CONDITIONS: Acute Myelogenous Leukemia; AML; Acute Myeloid Leukemia
Keywords: GDC-0199; Acute Myelogenous Leukemia; AML; ABT-199; Acute Myeloid Leukemia; Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-199 (Experimental): Continuous dosing of venetoclax (ABT-199) QD (once daily) beginning with dose-escalation on Week 1 Day 1. Participants received a dose of 20 mg of ABT-199 on Week 1 Day 1, 50 mg on Day 2, 100 mg on Day 3, 200 mg on Day 4, 400 mg on Day 5, 800 mg on Day 6 and QD thereafter.
  Interventions: Drug: ABT-199

INTERVENTIONS:
Drug: ABT-199 — Tablet
  Other Names: ABT-199 also known as venetoclax

SUMMARY:
This was a Phase 2, open-label, multicenter study evaluating the preliminary efficacy and safety of venetoclax (ABT-199) administered orally in participants with acute myelogenous leukemia (AML).

DETAILED DESCRIPTION:
The primary objective was to evaluate the preliminary efficacy of venetoclax administered orally in participants with relapsed and/or refractory (R/R) acute myelogenous leukemia (AML) or frontline therapy in patients with AML who were unfit for intensive therapy. The secondary objective was to evaluate the preliminary safety of venetoclax administered orally in patients with AML. The first portion of the study was to consist of 19 participants with the objective of evaluating anti-tumor effects and confirming the safety of the regimen. The second portion (expansion) was to consist of 35 additional subjects to evaluate anti-tumor effects and safety and was to commence if an adequate efficacy signal (i.e., ≥ 5/19 achieved complete remission [CR], CR with incomplete bone marrow recovery [CRi] or partial remission [PR]) had been observed in the first portion of the study. The criterion for success would have been met if ≥ 16 of 54 participants achieved remission. The efficacy signal from first portion of the study was deemed insufficient for enrollment into the second portion of the study, as 4 of the 19 subjects achieved CR/CRi. During the trial, a number of participants were in screening at the point of the interim analysis. Given the early signs of clinical activity of venetoclax, disease severity, and prognosis of these participants without available options for therapy, they were allowed to initiate treatment ahead of completion of the interim analysis. Therefore, 32 participants were enrolled. No additional participants were screened or treated after the interim analysis was completed.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of relapsed or refractory acute myelogenous leukemia (AML) (by World Health Organization [WHO] classification) or untreated AML in participants who are unfit for intensive therapy.
2. Participant has an Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
3. Participant must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 50 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula using ideal body mass (IBM) instead of mass.
4. Participant must have adequate liver function as demonstrated by:

   * aspartate aminotransferase (AST) ≤ 3.0 × upper limit of normal (ULN)*
   * alanine aminotransferase (ALT) ≤ 3.0 × ULN*
   * bilirubin ≤ 1.5 × ULN* *unless considered due to leukemic organ involvement. (Participants with Gilbert's Syndrome may have had a bilirubin > 1.5 × ULN per discussion between the investigator and AbbVie medical monitor)

Exclusion Criteria:

1. Participant has received acute anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal or any investigational therapy within 14 days or 5 half-lives (whichever is shorter) prior to first dose of ABT-199.
2. Participant has received a monoclonal antibody for anti-neoplastic intent within 8 weeks prior to the first dose of study drug.
3. Participant has received potent Cytochrome P450, family 3, subfamily A (CYP3A) inducers (such as rifampin, carbamazepine, phenytoin and St. John's wort) and warfarin or requires the use of warfarin (due to potential drug-drug interactions that may potentially increase the exposure of warfarin and complications of this effect) within 7 days prior to the first dose of study drug.
4. Participant has received CYP3A inhibitors (such as fluconazole, ketoconazole, and clarithromycin) within 5 days prior to the first dose of study drug.
5. Participant has a white blood cell count > 25 x 10^9/L.
6. Participant has acute promyelocytic leukemia (French-American-British Class M3 AML).
7. Participants with known active central nervous system (CNS) disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jalaja Potluri, MD, Study Director — AbbVie

REFERENCES:
- [Result] Konopleva M, Pollyea DA, Potluri J, Chyla B, Hogdal L, Busman T, McKeegan E, Salem AH, Zhu M, Ricker JL, Blum W, DiNardo CD, Kadia T, Dunbar M, Kirby R, Falotico N, Leverson J, Humerickhouse R, Mabry M, Stone R, Kantarjian H, Letai A. Efficacy and Biological Correlates of Response in a Phase II Study of Venetoclax Monotherapy in Patients with Acute Myelogenous Leukemia. Cancer Discov. 2016 Oct;6(10):1106-1117. doi: 10.1158/2159-8290.CD-16-0313. Epub 2016 Aug 12. PMID 27520294

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who received at least 1 dose of study drug
Period: Overall Study
Arm/Group | ABT-199
Started | 32
Treated | 32
Completed | 0
Not Completed | 32
Not completed — Progressive disease per protocol | 23
Not completed — Adv event related to progressive disease | 3
Not completed — Fatal progressive disease | 2
Not completed — Adverse event not related to progression | 1
Not completed — Chose palliative care | 1
Not completed — Proceeded to transplant | 1
Not completed — Removed from study due to no response | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Arm/Group | ABT-199
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Remission Rate
Description: The objective remission rate (ORR) was defined as the percentage of participants who achieved complete remission (CR), complete remission with incomplete bone marrow recovery (CRi), or partial remission (PR) per the International Working Group criteria for AML. Complete remission (CR) was defined as peripheral neutrophils at least 10˄3/μL, platelets ≥ 10˄5/μL and normocellular bone marrow with ≤ 5% blasts. Complete remission with incomplete bone marrow recovery (CRi) was defined as bone marrow with less than 5% blasts, with peripheral neutrophils of at least 10˄3/μL or platelets ≥ 10˄5/μL. Partial remission (PR) was defined as normalization in peripheral blood neutrophil and platelet counts with at least a 50% decrease in blasts persisting in bone marrow versus baseline.
Time Frame: When 19 participants had completed at least 12 weeks of treatment or after all enrolled participants had discontinued venetoclax, whichever was earlier
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-199
Number analyzed (Participants) | 32
percentage of participants | 18.8 [7.2 to 36.4]

2. Secondary Outcome: Complete Remission Rate
Description: The complete remission (CR) rate was defined as the percentage of participants who achieved CR per the International Working Group criteria for AML. Complete remission was defined as peripheral neutrophils at least 10˄3/μL, platelets ≥ 10˄5/μL and normocellular bone marrow with ≤ 5% blasts.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | ABT-199
Number analyzed (Participants) | 32
percentage of participants | 6.3

3. Secondary Outcome: Duration of Remission
Description: Duration of remission was defined as the number of days from the date of first remission (CR, CRi, or PR) per the International Working Group criteria for AML to the earliest recurrence or progressive disease (PD). In this study, the duration of remission analysis was not performed because of the low remission rate, per the Statistical Analysis Plan.
Time Frame: as for outcome 1
Population: The duration of remission analysis was not performed because of the low remission rate, per the Statistical Analysis Plan.
Arm/Group | ABT-199
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the number of months from the date of enrollment to the date of earliest disease progression. If a participant did not experience disease progression, then the data for that participant was censored at the date of the last disease assessment.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199
Number analyzed (Participants) | 32
months | 2.5 [1.0 to 3.0]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the number of months from the date of enrollment to the date of earliest progression or death. If a participant did not experience disease progression or death, then the data was censored at the date of the last disease assessment.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199
Number analyzed (Participants) | 32
months | 2.3 [1.0 to 2.7]

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the number of months from the date of enrollment to the date of death for all dosed participants. For participants who did not die, their data were censored at the date of last study visit or the last known date to be alive, whichever was later.
Time Frame: Measured up to 2 years after the last subject had enrolled in the study.
Population: All participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199
Number analyzed (Participants) | 32
months | 4.7 [2.3 to 6.0]

7. Secondary Outcome: Percentage of Participants Who Received Subsequent Stem Cell Transplant
Description: The percentage of participants who received a subsequent allogenic (from a healthy donor) stem cell transplant was summarized.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | ABT-199
Number analyzed (Participants) | 32
percentage of participants | 3.1

8. Secondary Outcome: Rate of Minimal Residual Disease (MRD) Negativity
Description: The rate of minimal residual disease (MRD) response was defined as the percentage of participants who had MRD negative status. Only participants with a reported MRD assessment (negative or positive) from the local laboratory at the investigator site were used in the calculation of MRD response rate.
Time Frame: as for outcome 1
Population: Participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-199
Number analyzed (Participants) | 23
percentage of participants | 43.5 [23.2 to 65.5]

9. Secondary Outcome: Complete Remission With Incomplete Marrow Recovery (CRi) Rate
Description: The complete remission with incomplete bone marrow recovery (CRi) rate was defined as the percentage of participants who achieved CRi per the International Working Group criteria for AML. Complete remission with incomplete bone marrow recovery was defined as bone marrow with less than 5% blasts, with peripheral neutrophils of at least 10˄3/μL or platelets ≥ 10˄5/μL.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | ABT-199
Number analyzed (Participants) | 32
percentage of participants | 12.5

10. Secondary Outcome: Complete Remission Rate and Complete Remission With Incomplete Marrow Recovery (CRi) Rate
Description: The complete remission rate and the complete remission with incomplete marrow recovery rate (Cri) was defined as the percentage of participants who achieved complete remission (CR) or complete remission with incomplete bone marrow recovery (CRi), per the International Working Group criteria for AML. Complete remission (CR) was defined as peripheral neutrophils at least 10˄3/μL, platelets ≥ 10˄5/μL and normocellular bone marrow with ≤ 5% blasts. Complete remission with incomplete bone marrow recovery (CRi) was defined as bone marrow with less than 5% blasts, with peripheral neutrophils of at least 10˄3/μL or platelets ≥ 10˄5/μL.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-199
Number analyzed (Participants) | 32
percentage of participants | 18.8 [7.2 to 36.4]

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time of study drug administration until 30 days after the last dose of study drug, up to 40 weeks.
Description: Serious adverse events occurring after the study-specific informed consent was signed but prior to the first dose of the investigational product were to be collected only if they were considered by the investigator to be causally related to the study required procedures.
Arm/Group | ABT-199
Serious Adverse Events (participants affected / at risk) | 27/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-199 (N=32)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 9
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
HYDROCELE (Congenital, familial and genetic disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
CROHN'S DISEASE (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
MESENTERITIS (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
DEATH (General disorders) | 1
PYREXIA (General disorders) | 1
BACTERAEMIA (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1
LEPTOTRICHIA INFECTION (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 5
PNEUMONIA FUNGAL (Infections and infestations) | 1
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1
PSEUDOMONAS INFECTION (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 2
SEPTIC SHOCK (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 2
VIRAL PHARYNGITIS (Infections and infestations) | 1
VULVAL CELLULITIS (Infections and infestations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
POST HERPETIC NEURALGIA (Nervous system disorders) | 1
PRESYNCOPE (Nervous system disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2
SCROTAL PAIN (Reproductive system and breast disorders) | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1
HYPOTENSION (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-199 (N=32)
ANAEMIA (Blood and lymphatic system disorders) | 4
ATRIAL FIBRILLATION (Cardiac disorders) | 3
SINUS BRADYCARDIA (Cardiac disorders) | 2
SINUS TACHYCARDIA (Cardiac disorders) | 4
EAR PAIN (Ear and labyrinth disorders) | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 7
CONSTIPATION (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 17
DYSPEPSIA (Gastrointestinal disorders) | 3
GINGIVAL BLEEDING (Gastrointestinal disorders) | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 19
STOMATITIS (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 13
ASTHENIA (General disorders) | 2
CHILLS (General disorders) | 2
FATIGUE (General disorders) | 11
MALAISE (General disorders) | 3
NON-CARDIAC CHEST PAIN (General disorders) | 4
OEDEMA PERIPHERAL (General disorders) | 8
PYREXIA (General disorders) | 6
CANDIDA INFECTION (Infections and infestations) | 2
CONJUNCTIVITIS (Infections and infestations) | 3
PNEUMONIA (Infections and infestations) | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
URINARY TRACT INFECTION (Infections and infestations) | 3
CONTUSION (Injury, poisoning and procedural complications) | 2
FALL (Injury, poisoning and procedural complications) | 3
LACERATION (Injury, poisoning and procedural complications) | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3
BLOOD BILIRUBIN INCREASED (Investigations) | 4
BLOOD CREATININE INCREASED (Investigations) | 2
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 2
WEIGHT DECREASED (Investigations) | 2
WEIGHT INCREASED (Investigations) | 2
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 4
FLUID OVERLOAD (Metabolism and nutrition disorders) | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 3
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 8
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 4
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 8
HYPOKALAEMIA (Metabolism and nutrition disorders) | 12
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 11
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
DIZZINESS (Nervous system disorders) | 2
DYSGEUSIA (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 11
SYNCOPE (Nervous system disorders) | 2
TREMOR (Nervous system disorders) | 2
ANXIETY (Psychiatric disorders) | 3
DELIRIUM (Psychiatric disorders) | 3
DEPRESSION (Psychiatric disorders) | 2
INSOMNIA (Psychiatric disorders) | 5
HAEMOGLOBINURIA (Renal and urinary disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 2
PURPURA (Skin and subcutaneous tissue disorders) | 2
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4
HYPERTENSION (Vascular disorders) | 4
HYPOTENSION (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.